CLINICAL TRIAL: NCT04970550
Title: Vaccination Against SARS-Cov2 in Chronic Inflammatory Rheumatism and Factors Determining Its Decision.
Brief Title: Vaccination Against SARS-Cov2 (COVID-19) in Chronic Inflammatory Rheumatism and Factors Determining Its Decision.
Acronym: VACCI-RIC
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01013-38
Record Dates: First submitted 2021-07-15; First posted 2021-07-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis
Keywords: SARS COV 2 vaccination
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non intervention — Non intervention

SUMMARY:
Rheumatoid arthritis and spondyloarthritis (ankylosing spondylitis and psoriatic arthritis mainly) are chronic inflammatory rheumatism (RIC), frequently onset in young adults. The prevalence is respectively 0.3 to 0.8% and 0.4%. or about 600,000 people. The "basic" treatments (DMARDs), essential to control the progression of the disease, are classified into csDMARDs (chemical), the first of which is methotrexate, or bDMARDs (biological). These treatments are immunomodulators and there is an increased risk of severe infection under these therapies. Several vaccinations are therefore recommended by learned societies in patients receiving these treatments, in order to prevent certain infectious risks.In the current pandemic context, the vaccination of these patients against SARS-Cov2 is a major issue in their management and is recommended by the French society of rheumatology. However, many patients express doubts about this vaccination or refuse it. The factors associated with the vaccination will are not known. Better identifying them would make it possible to adapt the information to be given to our patients to promote their adherence.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients
* Men or women of any age
* Follow-ups for chronic inflammatory rheumatism such as rheumatoid arthritis or spondyloarthritis
* Treated with methotrexate or biotherapy.

Exclusion Criteria:

* Patients not treated with biotherapy or methotrexate.
* Patients in whom the assessment could not be performed reliably

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A questionnaire is completed by the patient with the investigator during the medical consultation.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Determine the desire to be vaccinated against SARS-CoV2 | At inclusion
  Percentage of patients with RIC and treated with DMARDs who favor vaccination against SARS-CoV2 ; determined with a questionnaire

SECONDARY OUTCOMES:
Factors associated with the desire for vaccination against SARS-CoV2 | At inclusion
  Identify the factors associated with the desire for vaccination against SARS-CoV2 ; determined with a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: Undecided